CLINICAL TRIAL: NCT05206136
Title: Evaluation of Cervical and Lumbal Region Muscle Architecture in Individuals With Low Back and Neck Pain
Brief Title: Cervical and Lumbal Region Muscle Architecture in Individuals With Low Back and Neck Pain
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ozlem Ulger, Professor, Hacettepe University
Other Study IDs: GO 20/1034
Record Dates: First submitted 2022-01-07; First posted 2022-01-25 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Neck Pain; Back Pain
Keywords: neck pain; back pain; muscle architecture
MeSH Terms: conditions — Neck Pain; Back Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neck Pain Group: Patients with neck pain
  Interventions: Device: Ultrasonography
- Low Back Pain Group: Patients with low back pain
  Interventions: Device: Ultrasonography
- Healthy Individuals: Patients with no pain in neck or low back region
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Neck and Low back muscles will be evaluated by ultrasound.

SUMMARY:
Back or neck problems often begin with an injury and often include a muscle injury. Injury of muscle fibers can occur due to trauma, disease, myotoxic agents, inflammatory processes, and intense exercise. The level of muscle injury in low back or neck problems is unknown. However, the relationship between muscle injury and pain has been studied intensively.

Injury to skeletal muscles occurs when muscle activation begins abruptly and rapidly with muscle lengthening. Muscle pain that occurs with eccentric exercise peaks 24-48 hours after the exercise. Studies on this subject have generally focused on muscle fatigue, changes in the physiological structure of the muscle, and which muscle fiber types are injured more. Experimental studies focused on the results of skeletal muscle injury with early activation of the muscle during eccentric exercises. For example, it has been shown that mechanical changes in the tibialis anterior muscle occur in the first 5-7 minutes of exercise during eccentric exercise. Studies on the back and neck muscles are rare, and it has been stated that fatigue in these muscles plays an active role in the mechanism of injury. It is very difficult to accept this view directly, because there are different types of muscle fibers in the lower back and neck muscles. In terms of low back and neck pain and muscle injury, specific studies on muscle fiber types are required. In addition, muscle strength together with pain can change the load distribution to anatomical structures. However, muscle activity alters spinal stability and kinematics. It has been found that the M. Sternocleideomasteideus (M.SCM) muscle shows 5%-10% elongation tension during muscle activation, along with retraction in whiplash injuries. In deep muscle groups, this rate varies between 10% and 20%. It is not known to what extent the architectural features of the muscle change with these muscle tensions and to what extent the injury occurs when active extension occurs. It is clear that the relationship between muscle pain and injury should be examined in terms of biomechanical modeling, muscle architecture and outcomes.

Muscle length, fiber length, pennation angle, and physiological cross-sectional area (PCSA) values of many muscle groups, primarily the M.SCM and M.Transversus Abdominus muscles, were analyzed in healthy individuals. However, it is not known how it changes in individuals with low back or neck pain. For this reason, if the architectural features of the cervical and lumbar region muscles can be determined, since they are the muscles that are most affected by low back and neck problems and then exercised the most by physiotherapists, the relationship between injury and pain can be examined and correct muscle function can be achieved. The emergence of different values from healthy muscle architecture will be valuable in terms of correct exercise planning and proper function in individuals with low back and neck problems. The aim of working with this idea is to evaluate the architectural features of the cervical and lumbar region muscles in individuals with problems characterized by low back and neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neck or low back pain
* Healthy Individuals
* Between the ages of 18-60,
* Being literate,

Exclusion Criteria:

* Cervical radiculopathy, thoracic outlet syndrome,
* Malignant condition,
* Having systemic diseases such as neurological, psychological, cardiovascular and loss of function due to these diseases,
* A history of surgery in the spine and upper extremity, including the cervical region, in the last 1 year period,
* Fracture in the spine and upper extremity, including the cervical region, with a history of inflammation,
* Acute infection,
* Continuing another rehabilitation program,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with neck or low back pain and healthy individuals will be included in to study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of Neck and Low Back Muscle Thickness or PCSA with Ultrasonography | 15 minutes, muscles will be evaluated once.
  Ultrasonography is used to evaluate the architectural properties of the muscle (thickness or PCSA) in chronic painful musculoskeletal problems such as neck-back pain. Muscle architecture measurements of neck and low back muscles with ultrasound will be evaluated in the resting position by the specialist radiology doctor who is blind to the results of the study using 3.5-10 MHz convex and linear probes (Soundcam Mobile Ultrasound Device).

SECONDARY OUTCOMES:
Evaluation of pain severity | 5 minutes, pain intensity will be evaluated once.
  Visual Analogue Scale (VAS) indicates the level of pain that the person is experiencing at the moment, marked with a vertical line on a plane. The pain felt by the person is marked as "0: I feel no pain", "10: I feel very severe pain". Scoring is based on measuring the participant's vertical marking for pain on the plane with a ruler. The validity and reliability study of the scale was conducted by Price et al.
Evaluation of disability | 5 minutes, disability level will be evaluated once.
  Neck Disability Index (NDI) Vernon et al. developed by. The Turkish version study was conducted by Aslan et al. Made by. The NDI includes a total of 10 questions such as pain, personal care, concentration, working, driving, sleeping. Each question is scored between 0-5 points. 0 points means no restrictions, 50 points means complete apology. 0-4 points are evaluated as no disability, 5-14 points as mild disability, 14-24 points as moderate disability, 25-34 serious disability and 35 and above as complete disability.
  Oswestry Index (ODI) Fairbank et al. developed by. Questionnaire examines perceived level of disability in 10 everyday activities of daily living. For each section the total possible score is 5: if the first statement is marked the section score = 0; if the last statement is marked, 0-20%: Minimal disability,21-40%: Moderate Disability,41-60%: Severe Disability,61-80%: Crippling back pain,81-100%: Patients are either bed-bound or have an exaggeration of their symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dilara ONAN, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided